CLINICAL TRIAL: NCT04838821
Title: Randomized, Placebo-controlled, Double-blind, Multicenter Clinical Study to Compare the Efficacy and Safety of the Administration of Three Different Doses of an Anti-SARS-CoV-2 Hyperimmune Equine Serum Formulation in Hospitalized COVID-19 Patients (SECR-02)
Brief Title: Efficacy and Safety of Three Different Doses of an Anti SARS-CoV-2 Hyperimmune Equine Serum in COVID-19 Patients
Acronym: SECR-02
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Caja Costarricense de Seguro Social (Other Government)
Collaborators: Universidad de Costa Rica (Other); Ministry of Health Costa Rica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R020-SABI-00268
Record Dates: First submitted 2021-03-23; First posted 2021-04-09 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Covid19; Anti-SARS-CoV-2 hyperimmune equine serum; Neutralizing antibodies; Passive Immunotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 156 participants will be allocated randomly to either one of three treatment groups or to placebo through an internet based randomizer (Studyrandomizer.com). Participants can withdraw from the study at any time.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti SARS-CoV-2 equine hyperimmune serum (Experimental): All participants in the treatment groups will receive a single intravenous infusion on day 1 containing the specified dose according to their assigned group 12mg/kg, 30 mg/kg or 56mg/kg. Total volume of the infusion is 180ml, to be administered during a time period of at least 1 hour. Study participants will be followed during their hospitalization until they are discharged and on Study Day 28.
  Interventions: Biological: Anti SARS-CoV-2 equine hyperimmune serum
- Placebo (Experimental): All participants in the placebo group will receive a single intravenous infusion on day 1 containing a specified volume of a saline IV solution preparation. Total volume of the infusion is 180ml, to be administered during a time period of at least 1 hour. Study participants will be followed during their hospitalization until they are discharged and on Study Day 28.
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Anti SARS-CoV-2 equine hyperimmune serum — All participants in the treatment groups will receive a single intravenous infusion on day 1 containing the specified dose according to their assigned group 12mg/kg, 30 mg/kg or 56mg/kg. Total volume of the infusion is 180ml, to be administered during a time period of at least 1 hour. Study participants will be followed during their hospitalization until they are discharged and on Study Day 28.
  Arms: Anti SARS-CoV-2 equine hyperimmune serum
Biological: placebo — All participants in the placebo group will receive a single intravenous infusion on day 1 containing a specified volume of a saline IV solution preparation. Total volume of the infusion is 180ml, to be administered during a time period of at least 1 hour. Study participants will be followed during their hospitalization until they are discharged and on Study Day 28.
  Arms: Placebo

SUMMARY:
Passive immunotherapy is a therapeutic alternative used in a variety of infectious diseases including COVID-19. Equine polyclonal hyperimmune sera is a source of neutralizing antibodies against SARS-CoV-2 and a therapeutic alternative under investigation in COVID-19 patients. In the previous study NCT04610502 no significant variations were observed regarding efficacy and safety between two different pharmaceutical preparations of equine hyperimmune sera and adequate tolerability was reported with both investigational products. Formulations were produced through repeated immunization with viral recombinant proteins and contain either antibodies against SARS-CoV-2 S1 protein (S type) or a combination of viral proteins that included S1, N (nuclear), E (envelop) and M (membrane) (M type). Another investigation (NCT04494984) found that the administration of a pharmaceutical preparation similar to the S type produced clinical improvement in hospitalized patients with SARS-CoV-2 pneumonia, particularly those with severe disease.

Aim: Evaluate the efficacy and safety of three different doses of an anti-SARS-CoV-2 hyperimmune equine serum formulation (S-type) as an addition to the standard therapeutic approach in adult hospitalized patients with a diagnosis of moderate or severe COVID-19, radiological findings consistent with pneumonia and a symptom onset period not exceeding 10 days.

A total of 156 patients will be included and randomly divided into four groups, each group will receive a different dose of the investigational drug. On day 1, all participants will receive a single intravenous infusion containing the specified dose according to their assigned group. Clinical assessments, laboratory determinations that include: viral load, antibodies quantification, inflammatory and coagulation markers, cytokines levels as well as standard evaluations will be performed for each patient. Data will be collected for all groups on Days 0 to 7, 14 and 28 or at discharge after completion of treatment. The study will end for each participant on the day of discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects male or female, aged 18 and over.
2. Acceptance to participate in the study by the signature of the informed consent by the subject or relative (if applicable).
3. SARS-CoV-2 infection confirmed by reverse transcriptase -polymerase chain reaction (RT-PCR).
4. SARS-CoV-2 pneumonia confirmed by chest X-ray.
5. Patients with moderate or severe disease clinical presentation of the disease that require hospitalization.
6. Being within 10 days of the initial COVID-19 related symptoms onset.
7. Admission in the participating center within a 24hour period.
8. Female patients of child-bearing age with a negative pregnancy test.

Exclusion Criteria:

1. COVID-19 patients that do not require hospitalization (outpatient setting).
2. Patients who are participating in other therapeutic clinical trials.
3. COVID-19 patients who have received convalescent plasma treatment.
4. Critical disease COVID- 19 patients (respiratory failure, septic shock, and/or multiple organ dysfunction, admission PaO2/FIO2 ratio < 100).
5. Previously snake bitten individuals that received any type of equine hyperimmune serum treatment.
6. History of an allergic reaction due to contact or exposure to horses.
7. Pregnant or breastfeeding women.
8. Patients who, at the investigator´s discretion, are not likely to comply with study indications and procedures.
9. Patients currently undergoing hemodialysis in a renal support program.
10. Individuals who were previously classified by their treating physicians (prior to the COVID-19 diagnosis), of having an unfavorable prognosis with a short lifespan due to a concomitant disease other than the study disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-07-29 (Estimated); Study Completion 2021-09-29 (Estimated)

PRIMARY OUTCOMES:
Crude Mortality in COVID-19 patients | day 7 and 28
  The primary endpoint will be the difference in the proportion of deaths from all causes at 7 and 28 days after the administration of the investigational product between the study groups.

SECONDARY OUTCOMES:
Mechanical ventilation assistance (MVA) | day 28
  Change in MVA requirement days between study groups at day 28.
Hospital stay | day 28
  Change in the overall in-hospital at day 28 stay between study groups.
Inflammatory markers IL6 | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Changes in IL-6 levels to be evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
Inflammatory markers CRP | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Change in CRP levels to be evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
Inflammatory markers Procalcitonin | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Change in procalcitonin levels to be evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
Inflammatory markers Ferritin | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Change in ferritin levels to be evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
Thrombotic markers PTT | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Changes in PTT levels to evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
Thrombotic markers PT | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Changes in PT levels to evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
Thrombotic markers D Dimer | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Changes in D Dimer levels to evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
Thrombotic markers Fibrinogen | Days 0, 1, 2, 3, 5, 7, and 14 or discharge
  Changes in Fibrinogen levels to evaluated at days 0, 1, 2, 3, 5, 7, 14 or at time of discharge between study groups.
SpO2/FIO2 ratio | Days 0, 1, 2, 3, 4, 5, 6, 7 and 14 or discharge
  Change in the SpO2/FIO2 ratio to evaluated at days 0, 1, 2, 3, 4, 5, 6, 7 and 14 or at time of discharge between study groups
Changes in viral load | Days 0, 3, 7
  Change in viral load from baseline to 3 and 7 days after the start of the treatment between study groups
Modified Sequential Organ Failure Assessment (mSOFA) | Time Frame: Days 0, 1, 2, 3, 5, 7 and 14 or discharge
  Change in the mSOFA score to evaluated at days 0, 1, 2, 3, 5, 7 and 14 or at time of discharge between study groups.
WHO 8 point ordinal scale | Days 0, 1, 2, 3, 4, 5, 6, 7, 14 and 28 or discharge
  Change in the WHO 8 point ordinal scale of clinical status to evaluated at days 0, 1, 2, 3, 4, 5, 6, 7, 14 and 28 or at time of discharge between study groups.
Anti SARS-CoV-2 antibodies | Days 0, 1, 2, 3, 5, 7 and 14 or discharge
  Change in the anti SARS-CoV-2 antibodies titer levels to evaluated at days 0, 1, 2, 3, 5, 7 and 14 or at time of discharge between study groups.
Adverse events | day 28
  Incidence of adverse events as measured by CTCAE v. 5.0 at day 28 between study groups.

CONTACTS AND LOCATIONS:
Locations (4):
- Costa Rica (4):
  - Centro Especializado de Atención COVID19 (CEACO), San José
  - Hospital Dr. Rafael Ángel Calderón Guardia, San José
  - Hospital México, San José
  - Hospital San Juan de Dios, San José

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimber C, Valk SJ, Chai KL, Piechotta V, Iannizzi C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Hyperimmune immunoglobulin for people with COVID-19. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD015167. doi: 10.1002/14651858.CD015167.pub2. PMID 36700518